CLINICAL TRIAL: NCT02177292
Title: A Phase II Trial of High-Dose Pelvic Lymph Node IMRT( Intensity Modulated Radiation Therapy) and Hypofractionated Prostate IMRT for High Risk Prostate Cancer Patients
Brief Title: High-Dose Lymph Node Intensity Modulated Radiation Therapy and Hypofractionated Prostate (SIB)
Acronym: SIB
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical College of Wisconsin (Other)
Responsible Party: Principal Investigator, William Hall, Professor, Medical College of Wisconsin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO00013374
Record Dates: First submitted 2014-06-18; First posted 2014-06-27 (Estimated); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy; Radiotherapy, Intensity-Modulated; Radiotherapy, Image-Guided

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- IMRT & IGRT Radiation Therapy (Experimental): In this study we will deliver a high dose of radiation to the pelvic lymph nodes of 56 Gy (Gy/Gray = measure of amount of radiation) and at the same time give a boost (additional) radiation to the prostate itself (to 70 Gy).
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — A high dose of radiation to the pelvic lymph nodes of 56 Gy (Gy/Gray = measure of amount of radiation) and at the same time give a boost (additional) radiation to the prostate itself (to 70 Gy).
  Other Names: Intensity Modulated Radiation Therapy (IMRT) and Image Guided Radiation Therapy (IGRT).

SUMMARY:
The purpose of this study is to find out the effects (good and bad) of using newer technologies that allow very precise delivery of radiation. These newer technologies are Intensity Modulated Radiation Therapy (IMRT) and Image Guided Radiation Therapy (IGRT).

DETAILED DESCRIPTION:
In this study the treating physicians will deliver a high dose of radiation to pelvic lymph nodes of 56 Gy (Gy/Gray = measure of amount of radiation) and at the same time give a boost (additional) radiation to the prostate itself (to 70 Gy). The study will evaluate the response of the cancer and side effects of radiation to pelvic lymph nodes and to the prostate.

It is hoped that these newer technologies will:

1. allow a higher daily dose of radiation to the tumor and pelvic nodes
2. avoid nearby normal tissue and organs like the rectum and bladder
3. prevent the cancer from spreading or coming back

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, adenocarcinoma of the prostate
* T1-2N0M0 with risk of pelvic lymph nodes involvement >25% by Roach formula [(2/3xPSA) + (Gleason Score - 6)x10], or any T3-4N0M0
* Karnofsky Performance Scale > 70.
* Prostate tumor biopsy grading by Gleason score classification is mandatory prior to registration.
* No prior pelvic or prostate radiation or chemotherapy for any reason; induction hormonal therapy prior to registration is acceptable.
* Patients must sign a study-specific consent form prior to registration.
* No evidence of distant metastases (Bone scanning)

Exclusion Criteria:

* Clinical or pathological evidence of distant metastases (M1).
* Radical surgery for carcinoma of the prostate
* History of prior chemotherapy
* History of prior pelvic radiation therapy
* Children (age < 18).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2010-06-23 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2030-06-21 (Estimated)

PRIMARY OUTCOMES:
Change from baseline PSA level | 4 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 7 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 10 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 13 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 16 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 19 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 22 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 25 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 31 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 37 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 43 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 49 months
  PSA level in blood is measured in units of nanograms per milliliter.
Change from baseline PSA level | 55 months
  PSA level in blood is measured in units of nanograms per milliliter.

CONTACTS AND LOCATIONS:
Overall Officials: William Hall, MD, Principal Investigator — Medical College of Wisconsin
Locations (1):
- Froedtert & the Medical College of Wisconsin, Milwaukee, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kupelian PA, Willoughby TR, Reddy CA, Klein EA, Mahadevan A. Hypofractionated intensity-modulated radiotherapy (70 Gy at 2.5 Gy per fraction) for localized prostate cancer: Cleveland Clinic experience. Int J Radiat Oncol Biol Phys. 2007 Aug 1;68(5):1424-30. doi: 10.1016/j.ijrobp.2007.01.067. Epub 2007 Jun 4. PMID 17544601